CLINICAL TRIAL: NCT07309042
Title: A Randomized, Open-label Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics of the Combination of YN001 and Oral Rosuvastatin Calcium Tablets in Healthy Chinese Individuals
Brief Title: Phase 1 Study of the Safety and Pharmacokinetics of YN001 With Rosuvastatin in Healthy Chinese Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YN001-105
Record Dates: First submitted 2025-11-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerotic Cardiovascular Diseases; Cerebrovascular Diseases
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YN001 (Other)
  Interventions: Drug: YN001, Rosuvastatin calcium Tablets
- YN001+ Rosuvastatin calcium Tablets (Other)
  Interventions: Drug: YN001, Rosuvastatin calcium Tablets
- Rosuvastatin calcium Tablets (Other)
  Interventions: Drug: YN001, Rosuvastatin calcium Tablets

INTERVENTIONS:
Drug: YN001, Rosuvastatin calcium Tablets — Cycle 1 (Day 1 to day 14) : YN001, 40 mg, once a week, intravenous infusion, administered on day 1 and day 8, for a total of 2 doses. Cycle 2 (days 22 to 35) : YN001, 40 mg, once a week, intravenous infusion, administration on days 22 and 29, for a total of two doses. Rosuvastatin calcium Tablets, 10 mg, once a night, orally. Cycle 3 (Days 43 to 56) : Rosuvastatin calcium Tablets, 10 mg, once a night, orally.
  Arms: YN001
Drug: YN001, Rosuvastatin calcium Tablets — Cycle 1 (Day 1 to day 14) : YN001, 40 mg, once a week, intravenous infusion, administered on day 1 and day 8, for a total of two doses. Rosuvastatin calcium Tablets, 10 mg, once a night, oral administration. Cycle 2 (Days 22 to 35) : Rosuvastatin calcium Tablets, 10 mg, once a night, orally. Cycle 3 (days 43 to 56) : YN001, 40 mg, once a week, intravenous infusion, administration of D43 and D50, for a total of two doses.
  Arms: YN001+ Rosuvastatin calcium Tablets
Drug: YN001, Rosuvastatin calcium Tablets — Cycle 1 (Day 1 to day 14) : Rosuvastatin calcium Tablets, 10 mg, once a night, orally. Cycle 2 (Days 22 to 35) : YN001, 40 mg, once a week, intravenous infusion. Cycle 3 (days 43 to 56) : YN001, 40 mg, once a week, intravenous infusion, administration of D43 and D50, for a total of two doses. Rosuvastatin calcium Tablets, 10 mg, once a night, oral administration.
  Arms: Rosuvastatin calcium Tablets

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of YN001 in combination with rosuvastatin, so as to provide evidence for the feasibility of YN001 combined with statins in subsequent clinical trials.

DETAILED DESCRIPTION:
The primary objective of this study is to generate the evidence on the safety, tolerability and pharmacokinetic (PK) interaction profile of YN001 when combined with rosuvastatin, a widely prescribed high-intensity statin.

YN001 is being developed for patients with atherosclerotic cardiovascular disease (ASCVD) or at high cardiovascular risk. In these populations, contemporary treatment guidelines recommend statin therapy as foundational background treatment. However, because the human safety and PK profile of YN001 in combination with statins have not yet been established, concomitant statin use has been prohibited in all completed, ongoing, and planned YN001 clinical trials. This restriction creates a clinically and regulatorily important evidence gap: for YN001 to be used in its intended population, it is essential to determine whether co-administration with rosuvastatin is safe and whether either drug's systemic exposure is meaningfully altered.

To address this gap, the present study is designed as a single-centre, randomised, open-label, 3-sequence, 3-period crossover trial in healthy volunteers. The study will evaluate the the safety, tolerability and pharmacokinetics of repeated-dose intravenous YN001 administered alone and in combination with oral rosuvastatin calcium.

A total of 24 subjects will be enrolled. After screening, eligible participants will be randomly allocated 1:1:1 to three cohorts (8 per cohort, target 1:1 sex ratio). Each cohort will undergo three 14-day treatment periods separated by a 7-day wash-out (permissible window ±7 days).

The results of this study will inform whether concomitant statin can be safely permitted in subsequent Phase II and Phase III YN001 clinical trials, thereby enabling evaluation of YN001 in the intended ASCVD and high-cardiovascular-risk populations for whom chronic statin therapy is standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, characteristics, research methods and potential adverse reactions of this study, voluntarily participate in the study as a subject, and sign the Informed Consent Form (ICF) before any assessments are performed.
2. Healthy Chinese male and female subjects aged 18 to 55 years (inclusive, based on the age at the time of signing the ICF).
3. Body weight ≥ 50 kg for males and ≥ 45 kg for females; body mass index (BMI) ranging from 18 to 28 kg/m² (including the critical values).
4. Judged by the investigator based on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function) and viral serological test results (normal or abnormal without clinical significance) to be in good general health.
5. Female subjects must be non-pregnant and non-lactating; female subjects of childbearing potential (including female partners of male subjects) must agree to use effective contraceptive methods such as abstinence, condoms, intrauterine devices in use, double barrier methods (e.g., condoms plus diaphragms) from the screening period until 6 months after receiving the last dose of the study drug.
6. Willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Participation in other clinical trials within 3 months prior to the first dose or within 5 half-lives (whichever is longer). Subjects who withdrew from the study before receiving the study drug (i.e., not administered the drug) are eligible for enrollment.
2. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health supplements within 2 weeks prior to the first dose, or receipt of any type of vaccination.
3. Consumption of diets that may affect the in vivo metabolism of drugs (including grapefruit or grapefruit products, pitaya, mango, etc.) within 7 days prior to screening, engagement in strenuous exercise, or consumption of other diets that the investigator deems may affect the absorption, distribution, metabolism, or excretion of drugs.
4. History of severe food allergies (e.g., anaphylactic shock). Mild food allergies such as lactose intolerance and glucose intolerance are not excluded.
5. Allergy to multiple drugs, history of allergy to rosuvastatin, or history of allergic reactions to any component of the study drugs.
6. Known presence of clinically significant abnormal diseases or factors, including but not limited to clinically significant abnormalities in abdominal color Doppler ultrasound (liver, gallbladder, spleen, pancreas, bilateral kidneys, ureters, urinary bladder), chest posteroanterior radiography, etc.; or clinically significant diseases (including but not limited to diseases of the digestive system, circulatory system, respiratory system, endocrine system, urinary system, immune system, nervous system, and mental and psychological diseases) shown by other clinical findings within 6 months prior to screening.
7. History of myopathy/myalgia, or predisposition to myopathy/rhabdomyolysis (e.g., family history of hereditary myopathy, previous combined use of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors and fibrates, etc.).
8. Presence of hypothyroidism or hyperthyroidism.
9. History of acute or chronic bronchospastic diseases (including asthma, chronic obstructive pulmonary disease, whether treated or not) or heart failure, myocardial infarction, with a history of onset or recurrence within the past 3 years.
10. Known history of inflammatory bowel disease, ulcers, gastrointestinal bleeding, or rectal bleeding within 6 months prior to the first dose.
11. History of pancreatic injury or pancreatitis within 6 months prior to dosing.
12. Presence of symptoms of urinary tract obstruction or dysuria.
13. History of autonomic nervous system disorders (e.g., recurrent syncope, palpitations, etc.), with a history of onset or recurrence within the past 3 years.
14. Suffering from a major unhealed disease within 2 weeks prior to the first dose; or expected to undergo major surgery during the study period.
15. History of renal impairment, manifested by clinically significant abnormalities in creatinine, blood urea nitrogen (BUN) and/or urea levels, or clinically significant abnormalities in urine components (e.g., proteinuria).
16. Presence of liver disease or liver injury, or abnormal liver function test results. Subjects who meet any of the following criteria must be excluded from the study:

    1. Any one of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or serum bilirubin exceeds 1.5 times the upper limit of normal (ULN).
    2. Any two or more of ALT, AST, or serum bilirubin exceed the upper limit of normal (ULN).
17. History of clinically significant electrocardiogram (ECG) abnormalities; or presence of any of the following abnormalities during screening or baseline period:

    1. QTcF (males) > 470 milliseconds (msec).
    2. QTcF (females) > 480 milliseconds (msec). (Corrected by the Frederica formula, calculated as QTcF = QT/(RR⁰·³³))
18. Screening test shows hemoglobin level < 120 grams per liter (g/L) in males and < 110 grams per liter (g/L) in females.
19. Blood donation or blood loss exceeding 400 milliliters (mL) within 3 months prior to screening.
20. Smoking more than 10 cigarettes per day or habitual use of nicotine-containing products within 3 months prior to screening.
21. History of drug abuse within 12 months prior to screening; or use of any illegal drugs within 3 months prior to screening; or positive results in drug abuse tests (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, morphine, etc.) during screening.
22. Weekly alcohol consumption exceeding 14 standard drinking units (1 standard drinking unit = 285 mL of beer, or 25 mL of spirits, or 150 mL of wine) within 3 months prior to screening; or consumption of alcohol-containing products within 48 hours prior to the first dose; or positive results in breath alcohol test during the baseline period.
23. Positive results in tests for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum antibody.
24. The investigator deems the subject unsuitable for participation in the study due to any other diseases or conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 84 days

SECONDARY OUTCOMES:
Plasma pharmacokinetics: Maximum plasma concentration (Cmax) | 63 days
Number of Participants With ADA | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Chen, Master, Study Director — Beijing Inno Medicine Co., Ltd.

IPD SHARING:
Plan to Share IPD: No